CLINICAL TRIAL: NCT07077954
Title: COMPARISON OF THE EFFECTIVITY OF WARFARIN AND RIVAROXABAN IN THE TREATMENT OF LOWER LIMB DEEP VENOUS THROMBOSIS
Brief Title: COMPARISON OF WARFARIN AND RIVAROXABAN IN THE TREATMENT OF LOWER LIMB DEEP VENOUS THROMBOSIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children Hospital and Institute of Child Health, Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Adeel Ashiq, Senior Registrar, Children Hospital and Institute of Child Health, Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: adeel 8
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2023-07

CONDITIONS: Deep Vein Thrombosis (DVT)
Keywords: rivaroxaban; deep vein thrombosis; warfarin
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban given for DVT
  Interventions: Drug: Rivaroxaban
- Warfarin (Experimental): Warfarin given for DVT
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban used to treat DVT
  Arms: Rivaroxaban
Drug: Warfarin — warfarin used for DVT
  Arms: Warfarin

SUMMARY:
This was a randomized controlled trial conducted at General Surgical wards of Mayo Hospital, Lahore.Total 74(37 in each group) patients were included.After heparinizing patients for 48 hours (80 units/kg/stat and 18 units/kg/hour), patients in group-A were started Warfarin (5mg PO/OD), and patients in group-B received Rivaroxaban (15 mg PO/BD) for 21 days and then 20 mg PO/OD for 6 months. The dose of Warfarin was titrated according to INR (monitored on alternate days). Patients were discharged when limb girth was normal, as compared to opposite limb and pain was calmed. Length of stay was noted on day of discharge. Patient were followed on 6th and 12thweeks with doppler USGto assess the recanalization of all four segments including common femoral, superficial femoral, deep femoral and popliteal vein, percentage of recanalized segments was calculated out of total segments

DETAILED DESCRIPTION:
After approval from IRB, 74 patients meeting selection criteria were carefully chosen from all general surgical wards of Mayo Hospital. Informed written consent form was taken from all patients. Patients were randomized using lottery method and divided into two groups, A and B. History and clinical examination findings were noted. All baselines including INR was noted. USG Doppler findings documenting presence of thrombus in vein segments from common femoral to popliteal vein was noted. After heparinizing patients for 48 hours (80 units/kg stat and 18 units/kg per hour), patients in group A werestarted Warfarin (5mg PO OD), and patients in group B were given Rivaroxaban (15 mg PO BD) for 21 days and then 20 mg PO OD for 6 months. The dose of Warfarin was titrated according to INR (monitored on alternate days). While admitted in ward, monitoring was done for clinical improvement, including limb girth and pain severity.

Pain was assessed on scale of zero to 10, where 10 is most severe pain that patient ever had and zero is no pain at all. Limb girth was measured at mid-thigh, between greater trochanter and tibial tuberosity and compared to opposite limb and difference in limb girth was noted. Patients were discharged when limb girth was normal, as compared to opposite limb and pain was calmed. Length of stay was noted on day of discharge. Patient was kept on 6 weekly follow up till 12 weeks. Doppler USG was performed at 6 and 12 weeks to assess the recanalization of all four segments including common femoral, superficial femoral, deep femoral and popliteal vein, percentage of recanalized segments was calculated out of total segments at 6 and 12 weeks. Those patients, who were be able to come in person, were followed through telemedicine. All this data was recorded in proforma. After collection of data; length of stay and percentage of segments recanalized at 6 and 12 weeks were compared between groups.

Data Analysis Procedure Data was entered in SPSS v26.0. Quantitative variables including age and LOS was presented as Mean±SD. Qualitative variables including gender, vessel recanalization, was presented as frequency and percentages. Chi square test was applied to compare Recanalized segments between groups at 6th and 12th week post treatment respectively. Independent t-test was applied and p-value less than 0.05 was taken significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders aged between 16-70years presenting with clinical features (pain and swelling) of lower limb DVT, evidenced by USG Doppler. Thrombosis present in common femoral, superficial femoral, deep femoral and popliteal veins in one lower limb were included.

Exclusion Criteria:

* Exclusion Criteria: Patients taking other medications that can interact with warfarin or Rivaroxaban including aspirin, ibuprofen, clarithromycin, antihistamines, and SSRIs.Patients with co-morbid conditions that can affect coagulation, including CLD and CKD (CrCl<30), documented in previous hospital records. Pregnant and lactating females were excluded.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Recanalization | 12 weeks
  recanalization of all four segments including common femoral, superficial femoral, deep femoral and popliteal vein

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Adeel Ashiq, MBBS,MS, Principal Investigator — Children's Hospital, Lahore
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
As it is an intial study we will share after prolonged study